CLINICAL TRIAL: NCT01971970
Title: Biomarkers Predicting the Effect of Anti-TNF Treatment in Pediatric and Adult Inflammatory Bowel Disease
Brief Title: Biomarkers of Anti-TNF Treatment in Inflammatory Bowel Disease (IBD)
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, J.C. Escher, M.D., Ph.D, Associate Professor, Erasmus Medical Center
Other Study IDs: NL-42736.078.13
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Results first posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-11

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory bowel disease; Pediatric; Adult; Biomarker; Anti-TNF response; Infliximab; Adalimumab
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Infliximab; Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, gastrointestinal tract biopsies,buccal epithelium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric IBD patients: Anti-TNF naive patients with either Crohn's disease or ulcerative colitis will be treated with either Infliximab or Adalimumab
  Interventions: Biological: Infliximab; Biological: Adalimumab
- Adult IBD patients: Anti-TNF naive patients with either Crohn's disease or ulcerative colitis will be treated with either Infliximab or Adalimumab
  Interventions: Biological: Infliximab; Biological: Adalimumab

INTERVENTIONS:
Biological: Infliximab — Remission induction in anti-TNF naïve patients will be achieved by administration of 5 mg/kg IFX infusions at week 0, 2 and 6.
  Other Names: Remicade
Biological: Adalimumab — ADA is administered as subcutaneous injections every other week.In children (age below 18 years), remission induction in anti-TNF naïve patients will be achieved by an initial loading dose of 80 mg, followed by 40 mg 2 weeks later. In adults, remission is induced by 160 mg at week 0, followed by 80 mg at week 2
  Other Names: Humira

SUMMARY:
Anti-TNF treatment (infliximab (IFX), adalimumab (ADA)) has become standard therapy for refractory pediatric and adult Crohn's disease (CD) patients, and is used for the induction (primary response) and maintenance of remission. When effective, clinical and endoscopic remission is reached within weeks. However, primary non-response is observed in 20% of pediatric patients, and in 40% of adult CD patients, suggesting a more robust acute response to anti-TNF therapy in children as compared to adults.During maintenance treatment, 60 - 80% of patients have secondary loss of response, necessitating dose adjustments to maintain clinical response. Anti-TNF treatment is also increasingly used in ulcerative colitis (UC), and has been shown to induce remission in active disease. For UC, the comparison between the efficacy in children versus adults is more difficult to report as studies in children are scarce. Anti-TNF treatment is associated with rare but potentially fatal side effects, infusion reactions, and is an expensive treatment. To avoid overtreatment it is necessary to early identify non-responders to treatment, and therefore it is important to develop predictive biomarkers of treatment response.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a lifelong disease that may present during childhood in 20 - 25% of patients. There seems to be a worldwide trend towards increasing incidence rates of CD, especially in children. Patients with CD suffer from diarrhea, abdominal pain, nausea, malaise, and chronic malnutrition, in children often accompanied by growth failure and pubertal delay. CD is characterized by a transmural, granulomatous inflammation, involving any part of the gastrointestinal tract in a discontinuous manner.

Increased concentrations of tumor necrosis factor-α (TNFα) are found in the mucosa of CD patients , suggesting that TNF-α plays a pivotal role in the cytokine cascade of the inflammatory process. This key role of TNF-α has led to the development of biologic therapy based on the administration of monoclonal antibodies which bind and inactivate TNF-α. Infliximab (IFX, Remicade®) is a chimeric monoclonal antibody (75% human, 25% murine), while adalimumab (ADA, Humira®) is a fully human monoclonal antibody. Both antibodies bind with high affinity and specificity to soluble and membrane-bound TNF-α.

Anti-TNF drugs have become an important treatment strategy for CD patients who do not respond to or are intolerant of treatment with immunosuppressants (azathioprine, methotrexate) and corticosteroids. Anti-TNF induction therapy can induce complete clinical remission within weeks, often accompanied by mucosal healing. Interestingly, response to initial anti-TNF treatment is higher in pediatric CD patients (about 80%) than in adult CD patients (about 60%). Anti-TNF drugs do not cure CD: after their impressive initial effects, repeated infusions every 8 weeks or repeated subcutaneous injections every 2 weeks are necessary, while there is great concern about the long-term risks (infections, auto-immune disease, malignancy). Anti-TNF treatment is also increasingly used in ulcerative colitis, and has been shown to induce remission in active disease. For UC, the comparison between the efficacy in children versus adults is more difficult to report as studies in children are scarce. There are likely multiple host factors that influence the inter-individual variation in initial treatment response, such as disease phenotype, immune phenotype, and genetic background.

ELIGIBILITY:
Inclusion Criteria:

* Anti-TNF naïve CD patients (≥ 6 years) who initiate anti-TNF treatment (IFX or ADA) because of active luminal disease, failing treatment with immunomodulators (azathioprine, 6-mercaptopurine, methotrexate) and corticosteroids.
* Anti-TNF naïve UC patients (≥ 6 years) who initiate anti-TNF treatment (IFX or ADA) because of active disease despite corticosteroid treatment or because of failing of immunomodulator treatment.
* Anti-TNF naïve CD or UC patients (≥ 6 years) who initiate anti-TNF treatment (IFX or ADA) because of intolerance to treatment with immunomodulators (azathioprine, 6-mercaptopurine, methotrexate) or corticosteroids.
* Informed consent by patients and parents (when required).

Exclusion Criteria:

* IBD patients who initiate IFX or ADA immediately after diagnosis.
* Presence of severe perianal disease as primary indication to start anti-TNF treatment.
* Age < 6 years when anti-TNF maintenance treatment is initiated.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult IBD patients from the Department of Pediatric Gastroenterology of Erasmus MC-Sophia Children's Hospital and from the Department of Gastroenterology of Erasmus MC respectively.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10-30 (Actual); Study Completion 2017-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J C Escher, MD, PhD, Principal Investigator — Erasmus Medical Center - Sophia Children's Hospital; C J van der Woude, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Pediatric IBD Patients: Anti-TNF naive patients with either Crohn's disease or ulcerative colitis will be treated with either Infliximab or Adalimumab
  Infliximab: Remission induction in anti-TNF naïve patients will be achieved by administration of 5 mg/kg IFX infusions at week 0, 2 and 6.
  Adalimumab: ADA is administered as subcutaneous injections every other week.In children (age below 18 years), remission induction in anti-TNF naïve patients will be achieved by an initial loading dose of 80 mg, followed by 40 mg 2 weeks later.
- Adult IBD Patients: Anti-TNF naive patients with either Crohn's disease or ulcerative colitis will be treated with either Infliximab or Adalimumab
  Infliximab: Remission induction in anti-TNF naïve patients will be achieved by administration of 5 mg/kg IFX infusions at week 0, 2 and 6.
  Adalimumab: ADA is administered as subcutaneous injections every other week. In adults, remission is induced by 160 mg at week 0, followed by 80 mg at week 2
Period: Baseline Until Week 6
Arm/Group | Pediatric IBD Patients | Adult IBD Patients
Started | 24 | 21
Receiving Standard Therapy | 23 | 21
Therapy Escalation (Therapy escalation defined as either increasing anti-TNF dose or shortening interval between doses) | 1 | 0
Completed | 23 | 21
Not Completed | 1 | 0
Not completed — Stopped anti-TNF use | 1 | 0
Period: Week 6 Until Week 8
Arm/Group | Pediatric IBD Patients | Adult IBD Patients
Started | 23 | 21
Receiving Standard Therapy | 23 | 20
Completed | 23 | 20
Not Completed | 0 | 1
Not completed — Stopped anti-TNF use | 0 | 1
Period: Week 8 Until Week 14
Arm/Group | Pediatric IBD Patients | Adult IBD Patients
Started | 23 | 20
Receiving Standard Therapy | 16 | 19
Therapy Escalation (Therapy escalation defined as either increasing anti-TNF dose or shortening interval between doses) | 7 | 1
Completed | 23 | 20
Not Completed | 0 | 0
Period: Week 14 Until Week 22
Arm/Group | Pediatric IBD Patients | Adult IBD Patients
Started | 23 | 20
Receiving Standard Therapy | 12 | 16
Therapy Escalation (Therapy escalation defined as either increasing anti-TNF dose or shortening interval between doses) | 3 | 2
Completed | 23 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Week 22 Until Week 52
Arm/Group | Pediatric IBD Patients | Adult IBD Patients
Started | 23 | 19
Receiving Standard Therapy (Therapy escalation defined as either increasing anti-TNF dose or shortening interval between doses) | 5 | 9
Therapy Escalation (Therapy escalation defined as either increasing anti-TNF dose or shortening interval between doses) | 6 | 6
Completed | 15 | 15
Not Completed | 8 | 4
Not completed — Stopped anti-TNF use | 7 | 3
Not completed — Stopped anti-TNF use without escalation because of antibody-to-infliximab (ATI) formation | 1 | 0
Not completed — Stopped anti-TNF due to endoscopic improvement 1 year after start | 0 | 1
Period: Week 52 Until Week 78
Arm/Group | Pediatric IBD Patients | Adult IBD Patients
Started | 15 | 15
Completed | 14 | 12
Not Completed | 1 | 3
Not completed — Stopped anti-TNF use | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatric IBD Patients | Adult IBD Patients | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Age at Diagnosis | 13.24 [11.42 to 14.53] | 25.34 [19.53 to 35.65] | 15.47 [12.87 to 22.52]
  Age at start anti-TNF | 15.18 [12.79 to 15.76] | 33.46 [22.39 to 51.64] | 17.67 [15.17 to 31.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 12 | 11 | 23
Diagnosis Crohn's Disease [Count of Participants; unit: Participants] | 16 | 16 | 32
Disease Duration at start of anti-TNF [Median (Inter-Quartile Range); unit: years] | 1.025 [0.6 to 1.875] | 5.97 [2.37 to 10.42] | 1.69 [0.67 to 5.8]
Number of participants on Infliximab at start [Count of Participants; unit: Participants] | 23 | 18 | 41

OUTCOME MEASURES:

1. Primary Outcome: Pre-treatment Serum Level of Endogenous Anti-TNF in Relation to Primary Clinical Response or Non-response
Description: Pre-treatment serum level of endogenous anti-TNF are measured and analyzed in relation to primary clinical response or non-response
Time Frame: 8 weeks
Population: The pre-treatment serum levels of endogenous anti-TNF were zero in all 11 adult patients in whom endogenous anti-TNF was measured. Therefore, pre-treatment serum level of endogenous anti-TNF could not be fully analyzed in relation to primary clinical response or non-response.
Measure: Number; unit: endogenous anti-TNF serum level (µg/mL)
Arm/Group | Pediatric IBD Patients | Adult IBD Patients
Number analyzed (Participants) | 0 | 11
endogenous anti-TNF serum level (µg/mL) |  | NA — below the level of detection

2. Primary Outcome: RNA Expression Profiles in Relation to Clinical Endpoints
Description: Changes in week 0 and week 8 RNA expression profiles were evaluated in relation to the overall population and by study arm, i.e. either pediatric IBD or adult IBD.
Time Frame: 8 weeks
Population: Changes in week 0 and week 8 RNA expression profiles were analyzed within a subgroup of 29 patients (15 children and 14 adults) on infliximab treatment with samples taken at both week 0 and week 8. The number of genes with a 1.5 fold change (FDR value ≤ 0.05; paired t-test) from week 0 to week 8 were assessed for pediatric IBD or adult IBD patients.
Measure: Number; unit: Genes with 1.5 fold change (FDR value ≤
Units Other Than Participants: RNA expression profile samples
Groups:
- Overall: Overall combined data for pediatric and adult IBD patients
Arm/Group | Pediatric IBD Patients | Adult IBD Patients | Overall
Number analyzed (Participants) | 15 | 14 | 29
Number analyzed (RNA expression profile samples) | 15 | 14 | 29
Genes with 1.5 fold change (FDR value ≤ | 180 | 0 | 523
Statistical Analysis 1: Comparison: Pediatric IBD Patients vs Adult IBD Patients vs Overall; The number of genes with a 1.5 fold change (FDR value ≤ 0.05; paired t-test) from week 0 to week 8 were assessed for pediatric IBD or adult IBD patients; Test type: Equivalence — The number of genes with a 1.5 fold change (FDR value ≤ 0.05; paired t-test) from week 0 to week 8 were assessed for pediatric IBD or adult IBD patients; p < 0.05, Paired t-test,FDR 1.5fold,FDRvalue≤ 0.05

3. Secondary Outcome: Number of Participants With Clinical Endpoints of Interest.
Description: Clinical endpoints of Interest were the following:
  * Primary non-response was defined as no effect of anti-TNF after induction.
  * Remission and response were assessed at week 8 based on the appropriate disease activity scores for either children with Crohn's disease or ulcerative colitis (PCDAI and PUCAI respectively), or adults with Crohn's disease or ulcerative colitis (CDAI or Mayo score, respectively).
  * Continued use of anti-TNF was assessed 12 months and 18 months after start of anti-TNF.
Time Frame: Duration of study (start anti-TNF until 1 year after start of anti-TNF)
Measure: Count of Participants; unit: Participants
Groups:
- Adult IBD Patients: Anti-TNF naive patients with either Crohn's disease or ulcerative colitis will be treated with either Infliximab or Adalimumab
  Infliximab: Remission induction in anti-TNF naïve patients will be achieved by administration of 5 mg/kg IFX infusions at week 0, 2 and 6.
  Adalimumab: ADA is administered as subcutaneous injections every other week.In adults, remission is induced by 160 mg at week 0, followed by 80 mg at week 2
Arm/Group | Pediatric IBD Patients | Adult IBD Patients | Overall
Number analyzed (Participants) | 24 | 21 | 45
Participants
  Primary non-response | 1 | 1 | 2
  Remission at week 8 | 15 | 15 | 30
  Response at week 8 | 20 | 17 | 37
  Continued anti-TNF after 12 months | 15 | 15 | 30
  Continued anti-TNF after 18 months | 14 | 12 | 26
Statistical Analysis 1: Comparison: Pediatric IBD Patients vs Adult IBD Patients; Kaplan-Meier curves were produced by dividing the population in the following groups i) paediatric versus adult patients.These groups were used to statistically compare the proportions of patients over time regarding continued anti-TNF therapy, reflecting maintenance of response at 12 and 18 months; Test type: Other; p = 0.2616, gehan-breslow-wilcoxon test — Kaplan-Meier curve comparing the percentage of children and adults on continued anti-TNF therapy over the course of study duration

4. Secondary Outcome: Anti-TNF Treatment Specific Outcomes
Description: Anti-TNF treatment specific outcomes that were considered were:
  * Dose intensification; increase in dose of anti-TNF compared to standard therapy
  * Interval shortening; shortening of the interval of anti-TNFadministration compared to standard therapy.
  * Overall treatment intensification, the number of participants who underwent either dose intensification, interval shortening or both.
  * Development of Antibodies to infliximab during the course of follow-up
  * An infliximab serum trough level ≤ 3 mg/ml threshold (standard accepted therapeutic lower threshold) at week 14
Time Frame: Duration of study (start anti-TNF until 1 year after start of anti-TNF)
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric IBD Patients | Adult IBD Patients | Overall
Number analyzed (Participants) | 24 | 21 | 45
Participants
  Overall treatment intensification | 17 | 9 | 26
  Dose intensification | 14 | 4 | 18
  Interval shortening | 16 | 10 | 26
  Antibodies to infliximab Development | 4 | 3 | 7
  Infliximab serum trough level ≤ 3 mg/ml at week 14 | 7 | 4 | 11
Statistical Analysis 1: Comparison: Pediatric IBD Patients vs Adult IBD Patients; Kaplan-Meier curves were produced by dividing the population in the following groups i) paediatric versus adult patients.These groups were used to statistically compare the proportions of patients over time regarding the escalation of anti-TNF therapy (dose increase above 5 mg/kg and/or interval shortening to less than 8 weeks); Test type: Other; p = 0.0177, gehan-breslow-wilcoxon test — Kaplan-Meier curve comparing the percentage of children and adults with therapy intensification over the course of study duration

5. Secondary Outcome: Number of Participants With Concommitant Treatment
Description: Number of participants with concommitant treatment during the study was assessed. Concomitant treatment was defined as:
  * Additional use of immunomodulators such as methotrexate or azathioprine were registered.
  * Need for systemic prednisone, for instance in the case of an exacerbation, was assessed.
Time Frame: Duration of study (start anti-TNF until 1 year after start of anti-TNF)
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric IBD Patients | Adult IBD Patients | Overall
Number analyzed (Participants) | 24 | 21 | 45
Participants
  Addition of immunomodulators | 5 | 5 | 10
  Need for systemic prednisone | 3 | 0 | 3

ADVERSE EVENTS:
Arm/Group | Pediatric IBD Patients | Adult IBD Patients | Overall
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 0/45
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 0/45

LIMITATIONS AND CAVEATS:
Further analysis of clinical endpoints in relation to (clinical) biomarkers will be done by Mixed Model Analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No